CLINICAL TRIAL: NCT04458623
Title: Accuracy Of Air Test In Diagnosis Of Postoperative Lung Atelectasis In Elderly Patients Undergoing Major Orthopedic Surgery
Brief Title: Air Test In Diagnosis Of Postoperative Lung Atelectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasser Mamdouh Hassan Badawy, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: AOES
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- positive air test (Active Comparator): postoperative in the recovery room.patients received supplemental oxygen through a venture mask with a jet and flow adjusted to a theoretical fio2 of 100% for 10 min. The Air-Test was then performed by removing the oxygen mask and leaving the patients breathing room air for 10 min while continuously monitoring SpO2 with a pulse oximeter finger probe. The Air-Test result was considered positive when the recorded SpO2 was ≤96%.
  Interventions: Diagnostic Test: Air Test
- negative air test (Active Comparator): negative when SpO2 was >96 %.
  Interventions: Diagnostic Test: Air Test

INTERVENTIONS:
Diagnostic Test: Air Test — .The Air-Test may represent an accurate, simple, inexpensive and non-invasive method for diagnosing postoperative atelectasis.

SUMMARY:
Postoperative pulmonary complication represent asignificant source of morbidity and have greater incidence and costs than cardiac complications alone .Atelectasis is the commonest one. Aelectasis may develop in nearly up to 90% of patients after general anaesthesia ,persist up to several days .Oxygen therapy is usually given in the postoperative period to alleviate hypoxemia. However it's usually discontinued before discharge to the ward based on clinical criteria such as patients being awake with normal vital signs and no respiratory distress. Available literatures suggest that it's not valid . Pulse oximetry provide accurate objective measurement of oxygenation,continuous and non invasive.Recently, Fernando etal 2017,used pulse oximetry after 5 minutes of oxygenation to detect postoperative atelectasis, the cut point was 96%.

DETAILED DESCRIPTION:
Although it has been postulated that early hypoxemia lasts approximately two hours after a surgical procedure, the first 20 minutes of the postoperative period seem to be most critical . It is evident that the majority of transport times would fall well within this 20 minute window , thus the potential for postoperative hypoxemia during the transport period does exist. Canet, et al. (1989) found significant differences in oxygen saturation when administering 35% oxygen to adults in the PACU after a 30 second transport while breathing room air.The alveolar shunt induced by atelectasis is the main cause of oxygenation impairment during postoperative period. Witting MD, Lueck CH reported the ability of pulse oximetry at room air to detect hypoxemia based on 513 blood gas analysis. Coincidentially a room air oxygen saturation value <96% was selected a cut point of hypoxemia ( Po2 <70 mmhg )and moderate hypercapnia ( Pco2 >50 mmhg ) . Jones and Jones descriped a digram showing relationship between SPO2 and FiO2 and proved that SPO2 < 96% correspond to shunt effect of more than 10% and defines alveolar collapse . clark et al 2001determined time required for partial pressure of arterial oxygen to reach equilibrium during mechanical ventilation after a step change in fractional inspired oxygen, they reported that 5-10 minutes will be adequate . Ferrando C 2017 reported The accuracy of postoperative, non-invasive Air-Test to diagnose atelectasis in healthy patients after surgery They found that the air test diagnosed postoperative atelectasis with sensitivity of 82% and specificity of 87% and area uder the curve of 0.9 The presence of atelectasis was confirmed by CT scan in all patients with positive air test and in 5 patients with negative air test .The Air-Test may represent an accurate, simple, inexpensive and non-invasive method for diagnosing postoperative atelectasis.Sonography is a simple, noninvasive, and radiation-free methodology which has gained increasing usage in daily practice for detection of atelectasis. Sonography is a radiation-free methodology which plays an important role in diagnosing pulmonary diseases including obstructive and compressive atelectasis of different origins Furthermore, lung ultrasound has shown reliable sensitivity and specificity for the diagnosis of anaesthesia-induced atelectasis . Telectasis after general anaesthesia is basal and segmental. For this,we designed this trial as a pilot to detect the accuracy (sensitivity and specificity) of Air-Test to detect atelectasis in a homogenous group (elderly patients undergoing orthopedic surgery) using Roc testing.

ELIGIBILITY:
Inclusion Criteria:

* - Age (>60 years)
* ASA I , III
* Type of surgery: major orthopedic surgey

Exclusion Criteria:

* -Patient refusal.
* Patients with any significant chest disease
* Patients with any major cardiac disese
* Morbid obese

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
to assess the accuracy of air test in detecting postoperative atelectasis compared with reference ultrasonographic lung detection of atelectasis in a special grou of patients (aged) and a special form of surgery (orthopedics). | 30 minutes
  using air test

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine,Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleisher LA, Linde-Zwirble WT. Incidence, outcome, and attributable resource use associated with pulmonary and cardiac complications after major small and large bowel procedures. Perioper Med (Lond). 2014 Oct 7;3:7. doi: 10.1186/2047-0525-3-7. eCollection 2014. PMID 25313335
- [Background] Moller JT, Wittrup M, Johansen SH. Hypoxemia in the postanesthesia care unit: an observer study. Anesthesiology. 1990 Nov;73(5):890-5. doi: 10.1097/00000542-199011000-00016. PMID 2240679
- [Background] Brismar B, Hedenstierna G, Lundquist H, Strandberg A, Svensson L, Tokics L. Pulmonary densities during anesthesia with muscular relaxation--a proposal of atelectasis. Anesthesiology. 1985 Apr;62(4):422-8. doi: 10.1097/00000542-198504000-00009. PMID 3885791
- [Background] Canet J, Ricos M, Vidal F. Early postoperative arterial oxygen desaturation. Determining factors and response to oxygen therapy. Anesth Analg. 1989 Aug;69(2):207-12. PMID 2764289
- [Background] Jones JG, Jones SE. Discriminating between the effect of shunt and reduced VA/Q on arterial oxygen saturation is particularly useful in clinical practice. J Clin Monit Comput. 2000;16(5-6):337-50. doi: 10.1023/a:1011495416005. PMID 12580217
- [Background] Ferrando C, Romero C, Tusman G, Suarez-Sipmann F, Canet J, Dosda R, Valls P, Villena A, Serralta F, Jurado A, Carrizo J, Navarro J, Parrilla C, Romero JE, Pozo N, Soro M, Villar J, Belda FJ. The accuracy of postoperative, non-invasive Air-Test to diagnose atelectasis in healthy patients after surgery: a prospective, diagnostic pilot study. BMJ Open. 2017 May 29;7(5):e015560. doi: 10.1136/bmjopen-2016-015560. PMID 28554935
- [Background] Acosta CM, Maidana GA, Jacovitti D, Belaunzaran A, Cereceda S, Rae E, Molina A, Gonorazky S, Bohm SH, Tusman G. Accuracy of transthoracic lung ultrasound for diagnosing anesthesia-induced atelectasis in children. Anesthesiology. 2014 Jun;120(6):1370-9. doi: 10.1097/ALN.0000000000000231. PMID 24662376